CLINICAL TRIAL: NCT00316173
Title: An Open-Label, Single-Arm, Phase II Study of IV Weekly (Days 1 and 8 Every 21 Days) HYCAMTIN in Combination With Carboplatin (Day 1 Every 21 Days) as Second-Line Therapy in Subjects With Potentially Platinum-Sensitive Relapsed Ovarian Cancer
Brief Title: Second-Line Therapy Study For Potentially Platinum-Sensitive Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104864/902
Record Dates: First submitted 2006-04-19; First posted 2006-04-20 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Ovarian Cancer; Neoplasms, Ovarian
Keywords: HYCAMTIN; ovarian cancer; recurrent; relapsed; carboplatin; topotecan; potentially platinum-sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Topotecan; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm (Experimental): HYCAMTIN at a dose of 2.0 - 2.5mg/m2 on Days 1 and 8 every 21 days followed by carboplatin at AUC 5 on Day 1, every 21 days
  Interventions: Drug: topotecan; Drug: CARBOPLATIN

INTERVENTIONS:
Drug: topotecan — HYCAMTIN at a dose of 2.0 mg/m2 on Days 1 and 8 every 21 days followed by carboplatin at AUC 5 on Day 1
Drug: CARBOPLATIN — HYCAMTIN at a dose of 2.0 mg/m2 on Days 1 and 8 every 21 days followed by carboplatin at AUC 5 on Day 1

SUMMARY:
This study was designed to find the most effective and safest doses of both HYCAMTIN and CARBOPLATIN that can be given for the treatment of ovarian cancer. This study may allow researchers to determine the effectiveness of combining HYCAMTIN and CARBOPLATIN.

ELIGIBILITY:
Inclusion criteria:

* Subject must have baseline laboratory values as follows:
* Hemoglobin 9.0 g/dL
* Neutrophils 1,500/mm3
* Platelets 100,000/mm3
* Creatinine 1.5 mg/dL ( 133 mol/l) or creatinine clearance 60 mL/min
* Serum bilirubin < 2.0 mg/dL (< 35 umol/L)
* SGOT/AST, SGPT/ALT and alkaline phosphatase < 2 times ULN if liver metastases are absent by abdominal CT or MRI or < 5 times ULN if liver metastases are present
* Subject is allowed to have received, but is not required to have received, one additional prior non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition: Non-cytotoxic (biologic or cytostatic) agents include (but are not limited to) monoclonal antibodies, cytokines, and small-molecule inhibitors of signal transduction
* Subject is female 18 years of age with an ECOG Performance Status of 0, 1 or 2
* Subject has recurrent epithelial ovarian, fallopian tube, or primary peritoneal cancer which was histologically confirmed at the time of the primary diagnosis
* Subject has received one prior platinum-based chemotherapeutic regimen (containing either carboplatin or cisplatin) for the treatment of primary disease. Consolidation chemotherapy is not permitted
* Subject's disease is considered potentially platinum-sensitive (i.e., have had a platinum-free interval following complete response to carboplatin or cisplatin of greater than 6 months)
* Subject must have at least one measurable lesion as determined by diagnostic studies including CT or MRI or physical exam. Measurable disease must be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be 20 mm in their longest dimension when measured by conventional techniques, including palpation, plain X-ray, CT and MRI, or 10 mm when measured by spiral CT. Palpable tumor masses that cannot be evaluated radiologically must have 2 diameters 20 mm. An attempt to document lesion size by ultrasound should be undertaken for palpable lesions not visualized on CT (or MRI).
* The same diagnostic imaging method used to evaluate disease must be used throughout the study to evaluate lesions consistently
* Stable blood, liver and renal functions.
* Subjects of child-bearing potential must be practicing adequate contraception (e.g. oral contraceptives, diaphragm plus spermicide, or IUD) for at least 3 months prior to study start. The same contraceptive method should be used throughout the study and continue for at least 4 weeks after the end of the study

Exclusion criteria:

* Pregnant or lactating.
* Subject has received more than 1 prior chemotherapy regimen or a history of consolidation cytotoxic chemotherapy
* Subject has concomitant or history of previous malignancies, with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for 5 years
* Subject has brain metastases as documented by CT or MRI. Note: Asymptomatic subjects do not require CT or MRI to rule out brain metastases
* Received previous treatment with HYCAMTIN.
* Subject has received an investigational agent within 30 days or 5 half-lives (whichever is longer) prior to study entry
* Received prior radiation therapy for ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-03; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (18):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brightwaters, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Mayfield Heights, Ohio
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

REFERENCES:
- [Background] Rose PG, Monk BJ, Provencher D, Hartney J, Legenne P, Lane S. An open-label, single-arm Phase II study of intravenous weekly (Days 1 and 8) topotecan in combination with carboplatin (Day 1) every 21 days as second-line therapy in patients with platinum-sensitive relapsed ovarian cancer. Gynecol Oncol. 2011 Jan;120(1):38-42. doi: 10.1016/j.ygyno.2010.10.011. Epub 2010 Nov 5. PMID 21055798

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The run-in phase was conducted to find a safe dose of drug, before the treatment phase of the study began. Different doses were given to 22 participants (enrolled a few at a time) to find the safest dose. Once the safe dose was found, 55 new participants were enrolled in the treatment phase, and all were to start their treatment at this safe dose.
Groups:
- Dose-finding Phase: Starting dose of 2.0 milligrams (mg)/square meter (m2) topotecan (Days 1 and 8, every 21 days) and area under the curve (AUC) 5 carboplatin (Day 1 every 21 days)
- Activity Assessment Phase: Topotecan 2.5 mg/m2 (starting dose determined from the dose-finding phase) administered as a 30 minute intravenous (IV) infusion on Days 1 and 8, every 21 days. Carboplatin AUC 5 administered as a 30 minute IV infusion on Day 1, every 21 days.
Period: Run-in Phase
Arm/Group | Dose-finding Phase | Activity Assessment Phase
Started | 22 | 0
Completed | 15 | 0
Not Completed | 7 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Study Follow-up Stopped | 5 | 0
Period: Treatment Phase
Arm/Group | Dose-finding Phase | Activity Assessment Phase
Started | 0 | 55
Completed | 0 | 13
Not Completed | 0 | 42
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study Follow-up Stopped | 0 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-finding Phase | Activity Assessment Phase | Total
Number analyzed (Participants) | 22 | 55 | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.94) | 62.2 (11.13) | 62.6 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 55 | 77
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 2 | 2 | 4
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  White | 19 | 48 | 67
  Missing | 0 | 1 | 1
Number of participants with the indicated ECOG Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status assesses the effect of disease on daily living abilities, graded as: Grade 0: fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity; Grade 2: Capable of all selfcare, but unable to carry out any work activities.
  participants
    Grade 0 | 15 | 42 | 57
    Grade 1 | 7 | 9 | 16
    Grade 2 | 0 | 4 | 4

OUTCOME MEASURES:

1. Secondary Outcome: Time to Response
Description: Time to response was calculated as the time from start of treatment until first evidence of partial response (PR; >50% decrease in the measurements of the largest lesions with no appearance of new lesions) or complete response (CR; complete disappearance of all lesions).
Time Frame: From start of treatment to evidence of PR or CR (up to 39.3 weeks)
Population: All participants who showed a tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 17
weeks | 6.57 [5.86 to 12.57]

2. Secondary Outcome: Duration of Response
Description: Duration of response was calculated as the time from first documented PR or CR until disease progression or death. For participants who did not have disease progression or did not die, the date on which alternative anti-cancer therapy began was used, or the date of last contact (if sooner). The word used for such participants was "censored".
Time Frame: From time of PR or CR to disease progression/death (up to 56.0 weeks)
Population: All participants who showed a tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 17
weeks | 42.64 [36.14 to 47.14]

3. Primary Outcome: Number of Participants With the Indicated Response
Description: Overall response rate, as determined by radiologic evaluation (utilizing the World Health Organization [WHO] criteria and/or physical examination was measured. Complete response (CR: complete disappearance of all lesions), partial response (PR: >50% decrease in the measurements of the largest lesions with no appearance of new lesions), stable disease (SD: no change in tumor size for at least 8 weeks) and progressive disease (PD: >25% increase in measurements of lesions or appearance of new lesions).
Time Frame: From start of treatment to evidence of CR or PR (up to 39.3 weeks).
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 55
participants
  Complete response | 6
  Partial response | 11
  Stable disease | 20
  Progressive disease | 7
  Not evaluable | 11
Statistical Analysis 1: Comparison: Activity Assessment Phase; Test type: Superiority or Other; Percentage of participants with CR+PR = 30.9, 95% CI [18.7 to 43.1]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was calculated as the time from the start of treatment until disease progression or death. For participants who did not have disease progression or did not die, the date on which alternative anti-cancer therapy began was used, or the date of last contact (if sooner). The word used for such participants was "censored". Although "Time to Disease Progression" was stated as an endpoint in the protocol, the definition given in the protocol (and used in the study) was that of "PFS". As such, "PFS" was measured, not "Time to Disease Progression".
Time Frame: From start of treatment to disease progression/death (up to 67.7 weeks)
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 55
weeks | 44.29 [36.14 to 52.14]

5. Secondary Outcome: Number of Participants Who Died From the Start of Treatment to Follow-up
Description: The number of participants who died from the start of treatment to follow-up was calculated. For participants who did not die, the date of last contact was used. The word used for such participants was "censored".
Time Frame: From start of treatment to death (up to 110.4 weeks).
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 55
participants
  Died | 8
  Censored | 47

6. Secondary Outcome: The Number of Participants Classified as Responders in Cancer Antigen 125 (CA-125)
Description: CA-125 is a "tumor marker", found in greater concentration in tumor cells than other cells of the body. Participants were classed as responders if their CA-125 level at the end of study was 50% or less of baseline. In addition, a confirmatory sample (taken at least 28 days after the first sample) must have also been 50% or less of baseline.
Time Frame: Baseline to end of study (up to 54.7 weeks).
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 55
participants | 23

7. Secondary Outcome: Time to Disease Progression
Description: Although "Time to Disease Progression" was stated as an endpoint in the protocol, the definition given in the protocol (and used in the study) was that of "Progression-free Survival". As such, "Progression-free Survival" was measured, not "Time to Disease Progression". See the outcome measure entitled "Progression-free Survival" for data pertaining to time to disease progression.
Time Frame: From start of treatment to disease progression/death
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of study drug
Arm/Group | Activity Assessment Phase
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Adverse events that were rounded up to 5% in the CSR (e.g. 1/22; 4.54%) are also included here.
Arm/Group | Dose-finding Phase | Activity Assessment Phase
Serious Adverse Events (participants affected / at risk) | 6/22 | 12/55
Other Adverse Events (participants affected / at risk) | 20/22 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-finding Phase (N=22) | Activity Assessment Phase (N=55)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-finding Phase (N=22) | Activity Assessment Phase (N=55)
Fatigue (General disorders) | 14 | 42
Constipation (Gastrointestinal disorders) | 12 | 21
Nausea (Gastrointestinal disorders) | 10 | 40
Diarrhea (Gastrointestinal disorders) | 6 | 13
Anorexia (Metabolism and nutrition disorders) | 5 | 11
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Headache (Nervous system disorders) | 4 | 15
Dizziness (Nervous system disorders) | 4 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 16
Dysgeusia (Nervous system disorders) | 3 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 9
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Urinary tract infection (Infections and infestations) | 2 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 10
Insomnia (Psychiatric disorders) | 3 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Adverse drug reaction (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 9
Nasopharyngitis (Infections and infestations) | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Flushing (Vascular disorders) | 2 | 4
Drug hypersensitivity (Immune system disorders) | 2 | 12
Anemia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 4
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 5
Asthenia (General disorders) | 1 | 1
Catheter site related reaction (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Eye infection staphylococcal (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Anxiety (Psychiatric disorders) | 1 | 2
Libido decreased (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Atrial fibrillation (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Ear pruritis (Ear and labyrinth disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2
Urine abnormality (Renal and urinary disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Chest pain (General disorders) | 0 | 4
Mucosal inflammation (General disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 5
Pollakiuria (Renal and urinary disorders) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 3

LIMITATIONS AND CAVEATS:
As only 17 of 55 participants had CR/PR, the treatment was not effective. The follow up of participants for survival was thus stopped early (original plan: every 3 months for 2 years; then every 6 months for 3-5 years; then annually/until death).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.